CLINICAL TRIAL: NCT06133699
Title: A Prospective, Single-center, Clinical Trial to Evaluate the Efficacy of Sentinel Lymph Node Biopsy in Stage AI-IIA Germ Cell Tumors (Seminoma/Nonseminoma)(PITERLAND).
Brief Title: Sentinel Lymph Node Biopsy in Stage AI-IIA Germ Cell Tumors
Acronym: PITERLAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01112023-PITERLAND
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-11

CONDITIONS: Testicular Germ Cell Tumor
Keywords: testicular; Germ cell tumor; ICG; SLNB
MeSH Terms: conditions — Testicular Germ Cell Tumor; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SLNB (Experimental)
  Interventions: Procedure: Orchofuniculectomy with simultaneous laparoscopic biopsy of the sentinel lymph node using indocyanine green dye with/without methylene blue dye.; Diagnostic Test: Radiopharmaceutical administration (Technetium/methylene blue)

INTERVENTIONS:
Procedure: Orchofuniculectomy with simultaneous laparoscopic biopsy of the sentinel lymph node using indocyanine green dye with/without methylene blue dye. — Study participants will undergo orchofuniculectomy through an inguinal or laparoscopic approach. After completion of the orchofuniculectomy, indocyanine green (ICG) dye with or without methylene blue dye will be injected into the spermatic cord stump. Next step is detection with a gamma detector the sentinel lymph nodes and follow removing of one or more (up to 4) lymph nodes during laparoscopy. These lymph nodes will be sent for histological examination.
Diagnostic Test: Radiopharmaceutical administration (Technetium/methylene blue) — 24 hours before surgery, a radiotracer (RP) will be injected into the spermatic cord followed by SPECT to identify the regional sentinel lymph node(s).

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of sentinel lymph node biopsy in stage AI-IIA germ cell tumors (seminoma/nonseminoma). The main questions it aims to answer are:

* To evaluate relapse-free survival during the first two years after SLNB.
* To estimate the percentage of patients who did not require adjuvant treatment after primary endoscopic SLNB.
* Determine the microRNA expression profile in blood plasma, evaluate miRNAs as a potential prognostic and predictive factor in patients with testicular germ cell tumors.
* Assess the correlation between computed tomography and positive lymph nodes on examination.

Participants will undergo:

* surgical treatment including orchofuniculectomy with simultaneous laparoscopic biopsy of the sentinel lymph node using indocyanine green dye with/without methylene blue dye.
* 24 hours before the procedure, a radiopharmaceutical (RP) is injected into the spermatic cord, followed by SPECT to determine the regional sentinel lymph node(s).
* The level of microRNA will be examined before surgery and 10 days after surgery.

DETAILED DESCRIPTION:
Research Design This study is a prospective, single-center, non-randomized study evaluating the role of primary endoscopic SLNB on progression-free survival in patients with stage I-II germ cell seminoma/non-seminoma tumor without adjuvant treatment. Additionally, the study will determine the prognostic value of miRNAs as a noninvasive marker in clinical practice.

This study plans to recruit 44 male patients with a preliminary diagnosis of testicular tumor.

Patients who meet the inclusion/exclusion criteria will undergo surgical treatment including orchofuniculectomy with a simultaneous assessment and biopsy of the sentinel retroperitoneal lymph node.

The first stage of treatment Pre-operative preparation At the preoperative stage, it is planned to perform 3D modeling of computed tomography slices to visualize tumor conglomerates and vascular topography. A map of lymph node dissection zones will also be compiled. The anatomical boundaries of lymph node dissection are the aorta, the inferior vena cava, the iliac vessels, their bifurcation zones, the renal and mesenteric vessels. Due to the distribution of lymph nodes into cohorts (from 1 to 9 in each case), further histological examination of the surgical material will assess the completeness of the performed lymph node dissection.

Radiopharmaceutical administration (Technetium/methylene blue) 24 hours before surgery, a radiotracer (RP) will be injected into the spermatic cord followed by SPECT to identify the regional sentinel lymph node(s).

Orchofuniculectomy Study participants will undergo orchofuniculectomy through an inguinal or laparoscopic approach.

After completion of the orchofuniculectomy, indocyanine green (ICG) dye with or without methylene blue dye will be injected into the spermatic cord stump.

Second stage of treatment Laparoscopic access and port placement

Under general anesthesia, with the patient in the supine position with arms extended along the body and legs spread apart, after processing the surgical field, laparoscopic ports will be installed under sterile conditions as follows:

* In the pubic region, 1 cm below the navel, an optical trocar is installed according to the Hasson technique (pneumoperitoneum (P=14 mmHg).
* Installation of trocars in the right iliac region, in the left iliac region and above the pubic symphysis (5, 5 and 11 mm, respectively).

The patient is then placed in the Trendelenburg position. BSLU Next, in the operating room, the surgeon will use a gamma detector to determine the location of the sentinel lymph nodes, followed by removal of one or more (up to 4) lymph nodes from which the signal is received. These lymph nodes will be sent for histological examination.

The results of the work performed will present indicators of relapse-free survival after SLNB, as well as functional outcomes, such as postoperative complications, duration of hospital treatment, frequency of retrograde ejaculation in patients with stage IA-IIA testicular germ cell tumor. The data obtained will allow optimizing the selection of patients for surgical treatment, as well as identifying prognostic factors for the adjuvant stage of therapy.

Additionally, as part of the work, it is planned to study the expression profile of microRNAs in blood plasma, with subsequent assessment as a potential prognostic and predictive factor in patients with germ cell tumors. For this purpose, blood will be drawn from patients before surgery and 10 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male person at least 18 years of age at the time of signing the informed consent form;
* Provisional diagnosis of testicular tumor with isolated retroperitoneal lymphadenopathy;
* Computed tomography data of the abdominal cavity and retroperitoneal space with axial visualization of lymphadenopathy (within 6 weeks before the planned date of surgical treatment): at least one lymph node larger than 1 cm.

Exclusion Criteria:

* Severe or uncontrolled concomitant chronic diseases or acute diseases;
* Any condition that, in the opinion of the physician, may limit compliance with the study;
* Poor general condition (ECOG > 2, KPS < 70);
* Refusal of the patient to comply with the study procedures or refusal of the patient to continue participating in the study;
* Development of diseases or conditions that prevent the patient's continued participation in the study;
* AFP level is higher than reference values and / or b-hCG > 100 mIU/ml;
* Presence of a second malignant disease;
* History of systemic antitumor therapy and/or radiotherapy;
* Inadequate bone marrow, liver, kidney function: (Neutrophils < 1.5 x 10^9/l, Platelets < 100 x 10^9/l, ALT > 3 x ULN, AST > 3 x ULN, Total bilirubin > 1.5 xULN, GFR <35 ml/min)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival during the first two years after SLNB | two years
The percentage of patients who did not require adjuvant treatment after primary endoscopic SLNB | two years
Evaluation of miRNAs as a potential prognostic and prognostic factor in patients with testicular germ cell tumors. | two years
• Assess the correlation between computed tomography and positive lymph nodes on examination. | two years

SECONDARY OUTCOMES:
Сomplication rate | two years
All-cause mortality | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institute N.N. Petrov National Medical Research Center of Oncology Ministry of Health of the Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided